CLINICAL TRIAL: NCT03644615
Title: A Randomized Controlled Trial of a Mindfulness Program (MBSR) in the Management of Symptomatic Hip and Knee Osteoarthritis
Brief Title: A Mindfulness Program (MBSR) in the Management of Symptomatic Hip and Knee Osteoarthritis
Acronym: MINDFULNESS_OA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: RECHMPL17_0430; 2018-A00243-52 (Registry Identifier: ID-RCB)
Record Dates: First submitted 2018-08-21; First posted 2018-08-23 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2022-06

CONDITIONS: Osteoarthritis; Mindfulness; MBSR
Keywords: Osteoarthritis; Mindfulness; MBSR
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mindfluness and usual care (Experimental)
  Interventions: Other: Mindfluness and usual care
- Usual Care (Other)
  Interventions: Other: Usual care

INTERVENTIONS:
Other: Mindfluness and usual care — Intervention based on a mindfulness training program as a therapeutic alternative in osteoarthritis of the knee or hip. Mindfulness is a technique of attention training, which is to focus one's attention on the present moment and to examine the sensations that come to mind, how they appear, how they last time, and how they disappear.
  Arms: Mindfluness and usual care
Other: Usual care — No intervention on the patients
  Arms: Usual Care

SUMMARY:
Symptomatic osteoarthritis (OA) is the most common joint disease and the leading cause of disability in industrialized countries. Therapeutic approaches to prevent the development and progression of osteoarthritis are disappointing and very limited. New therapeutic alternatives seem essential to better manage his daily life. Non-drug approaches, including psycho-corporal approaches are increasingly used in the management of chronic pain.

Mindfulness is a technique of attention training, which is to focus one's attention on the present moment and to examine the sensations that come to mind, how they appear, how they last time, and how they disappear.

Regarding rheumatological pathologies, a Mindfulness Program (MBSR) has shown its effectiveness in chronic pain; and in particular in osteo-articular localization, such as chronic low back pain. A recent study found a correlation between a pre-disposition to mindfulness and less pain and / or better quality of life in patients with knee osteoarthritis. However, to the knowledge of investigator, no study has evaluated the effectiveness of an intervention based on a mindfulness training program as a therapeutic alternative in osteoarthritis of the knee or hip.

The goal of investigator is to evaluate, using a randomized, controlled study, the effect of a mindfulness program (according to the MBSR protocol) on pain, function, psychological state and quality of life patients with knee or hip osteoarthritis

ELIGIBILITY:
Inclusion Criteria:

* Osteoarthritis of the knee or hip (Kellgren and Lawrence X-ray stage ≥ 2)
* Mean pain VAS on at least one reference joint (knee or hip)> 40 mm during the last week
* Stable treatment with analgesics for at least a week

Exclusion Criteria:

* Corticosteroids (oral or injectable) in the month prior to inclusion
* Intra-articular injection of hyaluronic acid in the last 3 months prior to inclusion
* Inflammatory rheumatic disease (rheumatoid arthritis, spondyloarthritis, CCPD)
* Current depressive episode
* Psychotic disorders
* Usual practice of a relaxation method (mindfulness, yoga, sophrology ...)
* Major protected by law (guardianship, curatorship or under the safeguard of justice)
* Subject in a period of exclusion relative to another protocol or for which the annual amount maximum compensation of € 4500 has been reached.
* Subject participating in another research protocol
* Subject not affiliated to a social security
* Pregnant woman, parturient or nursing, patient unable to give her major consent protected, vulnerable persons (Articles L.1121-6, L.1121-7, L.1211-8, L.1211-9)
* Subject deprived of liberty by judicial or administrative decision

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-09-05 (Actual); Primary Completion 2019-03-04 (Actual); Study Completion 2019-09-04 (Actual)

PRIMARY OUTCOMES:
Evaluate the efficacy of a mindfulness program as a treatment for hip or knee osteoarthritis on the WOMAC pain score. | 6 months
  Improvement in WOMAC pain before and after the program in the MBSR group compared to control group. The WOMAC is a validated index in the assessment of lower extremity osteoarthritis, by the system of rating the answers to questions by a visual analogue scale from 0 to 100 mm. It is possible to calculate the scores in each domain (pain, stiffness and function) or for the whole WOMAC. This is a self-administered questionnaire completed by the patient.

SECONDARY OUTCOMES:
Changes in pain scores (VAS/100) between initiation visit and 3 months | 3 months
  EVA pain (visual analogue scale over 100 mm): one-dimensional measurement of the intensity of pain. EVA pain is a continuous scale consisting of a horizontal line from 0 (no pain) to 100 mm (maximum pain)
Changes in pain scores (VAS/100) between initiation visit and 6 months | 6 months
  EVA pain (visual analogue scale over 100 mm): one-dimensional measurement of the intensity of pain. EVA pain is a continuous scale consisting of a horizontal line from 0 (no pain) to 100 mm (maximum pain)
Changes in WOMAC questionnaire (total, pain, function and stiffness) between initiation visit and 3 months | 3 months
  The WOMAC is a validated index in the assessment of lower extremity osteoarthritis, by the system of rating the answers to questions by a visual analogue scale from 0 to 100 mm. It is possible to calculate the scores in each domain (pain, stiffness and function) or for the whole WOMAC. This is a self-administered questionnaire completed by the patient.
Changes in WOMAC questionnaire (total, pain, function and stiffness) between initiation visit and 6 months | 6 months
  The WOMAC is a validated index in the assessment of lower extremity osteoarthritis, by the system of rating the answers to questions by a visual analogue scale from 0 to 100 mm. It is possible to calculate the scores in each domain (pain, stiffness and function) or for the whole WOMAC. This is a self-administered questionnaire completed by the patient.
Changes in OARSI-OMERACT response criteria between initiation visit and 3 months | 3 months
  The responder rate is defined by an improvement of 20%, with an absolute variation ≥ 10mm, on 2 of the following 3 measures: WOMAC pain, WOMAC function and / or overall assessment of disease activity by the patient.
  The overall evaluation of the patient's disease activity is performed on a 100 mm horizontal visual analogue scale (0 = inactive disease, 100 = highly active disease). It is used for the global assessment of the activity of the disease by the patient.
Changes in OARSI-OMERACT response criteria between initiation visit and 6 months | 6 months
  The responder rate is defined by an improvement of 20%, with an absolute variation ≥ 10mm, on 2 of the following 3 measures: WOMAC pain, WOMAC function and / or overall assessment of disease activity by the patient.
  The overall evaluation of the patient's disease activity is performed on a 100 mm horizontal visual analogue scale (0 = inactive disease, 100 = highly active disease). It is used for the global assessment of the activity of the disease by the patient.
Changes in SF-36 score between initiation visit and 3 months | 3 months
  The SF-36 includes 36 items divided into 8 dimensions (physical functioning, limitations of functions related to physical health, physical pain, general health, vitality [energy / fatigue], functioning or social well-being, limitations of functions related to mental health, physical health) to which were added 4 items examining the cognitive functioning, from the "Medical Outcomes Study". This questionnaire was supplemented by questions aimed at clarifying the socio-demographic profile of the participants as well as the use of care services.
Changes in SF-36 score between initiation visit and 6 months | 6 months
  The SF-36 includes 36 items divided into 8 dimensions (physical functioning, limitations of functions related to physical health, physical pain, general health, vitality [energy / fatigue], functioning or social well-being, limitations of functions related to mental health, physical health) to which were added 4 items examining the cognitive functioning, from the "Medical Outcomes Study". This questionnaire was supplemented by questions aimed at clarifying the socio-demographic profile of the participants as well as the use of care services.
Changes in HAD score between initiation and 3 months | 3 months
  The Hospital Anxiety and Depression (HAD) questionnaire assesses the psychological impact of the patient. It consists of 14 questions with 4 possible answers. This score makes it possible to differentiate a level of anxiety and a level of depression according to the answers. Each sub-scale varies from 0 to 21
Changes in HAD score between initiation and 6 months | 6 months
  The Hospital Anxiety and Depression (HAD) questionnaire assesses the psychological impact of the patient. It consists of 14 questions with 4 possible answers. This score makes it possible to differentiate a level of anxiety and a level of depression according to the answers. Each sub-scale varies from 0 to 21

CONTACTS AND LOCATIONS:
Locations (1):
- Rhumatology Department - CHU Montpellier, Montpellier, France

REFERENCES:
- [Background] Marais C, Song Y, Ferreira R, Aounti S, Duflos C, Baptista G, Pers YM. Evaluation of mindfulness based stress reduction in symptomatic knee or hip osteoarthritis patients: a pilot randomized controlled trial. BMC Rheumatol. 2022 May 30;6(1):46. doi: 10.1186/s41927-022-00277-9. PMID 35637515
- See also: open access — https://rdcu.be/cODwx